CLINICAL TRIAL: NCT04411316
Title: Pharmacomechanical Catheter-directed Thrombolysis (PCDT) Plus Anticoagulation Compared to Anticoagulation Alone for Acute Primary Iliofemoral Deep Venous Thrombosis:
Brief Title: Catheter-directed Thrombolysis Compared to Anticoagulation Alone for Acute Primary Iliofemoral Deep Venous Thrombosis
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Zero Patients met criteria
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Principal Investigator, Ehab Eltahawy, MD, Associate professor of Medicine, University of Toledo Health Science Campus
Organization: University of Toledo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 300439
Record Dates: First submitted 2020-05-07; First posted 2020-06-02 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Deep Venous Thrombosis; Post Thrombotic Syndrome
MeSH Terms: conditions — Venous Thrombosis; Postthrombotic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Pharmacomechanical thrombolysis plus anticoagulation (Experimental): This group of patients will receive Pharmacomechanical catheter-directed thrombolysis (PCDT) plus Anticoagulation.
  PCDT will be AngioJet along with alteplase. Anticoagulation will be heparin only
  Interventions: Combination Product: Catheter directed thrombolysis plus anticoagulation
- Anticoagulation (Active Comparator): This group of patients will receive standard anticoagulation only. Anticoagulation will be Heparin only
  Interventions: Drug: Anticoagulation

INTERVENTIONS:
Combination Product: Catheter directed thrombolysis plus anticoagulation — Patients will be randomized to pharmacomechanical catheter directed thrombolysis plus anticoagulation.
  PCDT will be AngioJet along with alteplase.
  Other Names: Pharmacomechanical thrombolysis
  Arms: Pharmacomechanical thrombolysis plus anticoagulation
Drug: Anticoagulation — Patients will receive anticoagulation alone. Anticoagulation will be heparin only.
  Arms: Anticoagulation

SUMMARY:
Post-thrombotic syndrome (PTS) is a complication that can develop after deep vein thrombosis (DVT) of the lower extremities. PTS can occur at various times after the initial episode, but usually manifests within two years of initial DVT onset. Early and more complete thrombus clearance is believed by many to relieve venous outflow obstruction, preserve valvular function and reduce venous hypertension. Two previously published randomized controlled trials, the CAVENT trial and the ATTRACT trial, were larger and designed to investigate the efficacy of CDT. However, both of these trials included patients with iliofemoral as well as femoro-popliteal deep vein thrombosis. Our study will be limited to patients with iliofemoral deep vein thrombosis to assess whether Pharmacomechanical catheter-directed thrombolysis (PCDT) therapy utilizing AngioJet and tPA can safely and effectively reduce post thrombotic syndrome after 24 months.

DETAILED DESCRIPTION:
Patients with Iliofemoral DVT are theoretically at the highest risk for development of PRS given involvement of the major drainage pathway of both superficial femoral and deep femoral veins. This would not only affect the primary venous drainage, but would also compromise the ability to develop efficient collateral pathways. This creates higher chances of developing post-thrombotic syndrome (PTS). The proposed trial would utilize Angiojet thrombectomy followed by catheter directed thrombolysis and Anticoagulation compared to Anticoagulation alone. To assess whether Pharmacomechanical catheter-directed thrombolysis (PCDT) therapy utilizing AngioJet and tPA for the treatment of iliofemoral deep venous thrombosis can safely and effectively reduce post thrombotic syndrome after 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 and younger than 75
2. Symptomatic, proximal deep-vein thrombosis involving the Iliofemoral vein from 12/01/2019 to 12/01/2022

Exclusion Criteria:

1. Age less than 18 years or greater than 75 years.
2. Symptom duration > 14 days for the DVT episode in the index leg (i.e. non-acute DVT).
3. In the index leg: established PTS, or previous symptomatic DVT within the last 2 years.
4. In the contralateral (non-index) leg: symptomatic acute DVT a) involving the popliteal and/or tibial veins; or b) for which thrombolysis is planned as part of initial therapy.
5. Limb-threatening circulatory compromise.
6. PE with hemodynamic compromise (i.e. hypotension).
7. Inability to tolerate PCDT procedure due to severe dyspnea or acute systemic illness.
8. Allergy, hypersensitivity, or thrombocytopenia from heparin, rt-PA, or iodinated contrast, except for mild-moderate contrast allergies for which steroid pre-medication can be used.
9. Hemoglobin < 9.0 mg/dl, INR > 1.6 before warfarin was started, or platelets < 100,000 /ml.
10. Moderate renal impairment in diabetic patients (estimated GFR < 60 ml/min) or severe renal impairment in non-diabetic patients (estimated GFR < 30 ml/min).
11. Active bleeding, recent (< 3 months) GI bleeding, severe liver dysfunction, bleeding diathesis.
12. Recent (< 3 months) internal eye surgery or hemorrhagic retinopathy; recent (< 10 days) major surgery, cataract surgery, trauma, CPR, obstetrical delivery, or other invasive procedure.
13. History of stroke or intracranial/intraspinal bleed, tumor, vascular malformation, aneurysm.
14. Active cancer (metastatic, progressive, or treated within the last 6 months). Exception: patients with non-melanoma primary skin cancers are eligible to participate in the study.
15. Severe hypertension on repeated readings (systolic > 180mmHg or diastolic > 105 mmHg).
16. Pregnant (positive pregnancy test, women of childbearing potential must be tested).
17. Recently (< 2 years or chronic non-ambulatory status.
18. Use of a thienopryridine antiplatelet drug (except clopidogrel) in the last 5 days.
19. Life expectancy < 2 years or chronic non-ambulatory status.
20. Inability to provide informed consent or to comply with study assessments (e.g. due to cognitive impairment or geographic distance).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-12-19 (Estimated); Study Completion 2022-12-19 (Estimated)

PRIMARY OUTCOMES:
Post-thrombotic syndrome at any time between 6-month and 24-month. | 6-24 months
  Occurrence of post-thrombotic syndrome at any time between 6-month and 24-month after procedure by Villata score (Villata score >5 or more), or if patient underwent an unplanned endovascular procedure to treat venous symptoms.
  The variables in villata scores are pain, cramps, heaviness, parasthesia, pruritus, pretibial edema, skin induration, hyperpigmentation, pain during calf compression, venous ectasia and redness.
  The Villata score ranges 0-45. Villata score <5 means no post-thrombotic syndrome. Villata score 5-9 mild post-thrombotic syndrome. Villata score 10-14 means moderate post-thrombotic syndrome. Villata score ≥15 or presence of an ulcer indicates severe post-thrombotic syndrome.
  The more is the score the worse is the disease.

SECONDARY OUTCOMES:
Post-thrombotic syndrome at 6 months. | 6 months
  Occurrence of post-thrombotic syndrome at 6 months measured by Villata score (Villalta score was 5 or higher).
Post-thrombotic syndrome at 12 months. | 12 months
  Occurrence of post-thrombotic syndrome at 12 months measured by Villata score (Villalta score was 5 or higher).
Post-thrombotic syndrome at 18 months. | 18 months
  Occurrence of post-thrombotic syndrome at 18 months measured by Villata score (Villalta score was 5 or higher).
Post-thrombotic syndrome at 24 months. | 24 months
  Occurrence of post-thrombotic syndrome at 24 months measured by Villata score (Villalta score was 5 or higher).
Villalta scale at 6 months | 6 months
  The severity of the post-thrombotic syndrome to be evaluated at 6 months with the use of the Villalta scale
Villalta scale at 12 months | 12 months
  The severity of the post-thrombotic syndrome to be evaluated at 12 months with the use of the Villalta scale.
Villalta scale at 18 months | 18 months
  The severity of the post-thrombotic syndrome to be evaluated at 18 months with the use of the Villalta scale.
Villalta scale at 24 months | 24 months
  The severity of the post-thrombotic syndrome to be evaluated at 18 months with the use of the Villalta scale.
Venous Clinical Severity Score at 6 months | 6 months
  The severity of the post-thrombotic syndrome to be evaluated at 6 months with the use of the Venous Clinical Severity Score.
Venous Clinical Severity Score at 12 months | 12 months
  The severity of the post-thrombotic syndrome to be evaluated at 12 months with the use of the Venous Clinical Severity Score.
Venous Clinical Severity Score at 18 months | 18 months
  The severity of the post-thrombotic syndrome to be evaluated at 18 months with the use of the Venous Clinical Severity Score.
Venous Clinical Severity Score at 24 months | 24 months
  The severity of the post-thrombotic syndrome to be evaluated at 24 months with the use of the Venous Clinical Severity Score.
Health-Related Quality of Life AT 6 months | 6 months
  Health-Related Quality of Life measured by Venous Disease-Specific Quality of Life
Health-Related Quality of Life at 12 months. | 12 months
  Health-Related Quality of Life measured by Venous Disease-Specific Quality of Life at 12 months.
Health-Related Quality of Life at 18 months. | 18 months
  Health-Related Quality of Life measured by Venous Disease-Specific Quality of Life at 18 months.
Health-Related Quality of Life at 24 months. | 24 months
  Health-Related Quality of Life measured by Venous Disease-Specific Quality of Life at 24 months.
Health-Related Quality of Life at 6 months. | 6 months
  Health-Related Quality of Life measured by Generic Quality of Life at 6 months.
Health-Related Quality of Life at 12 months. | 12 months
  Health-Related Quality of Life measured by Generic Quality of Life at 12 months
Health-Related Quality of Life at 18 months. | 18 months
  Health-Related Quality of Life measured by Generic Quality of Life at 18 months.
Health-Related Quality of Life at 24 months. | 24 months
  Health-Related Quality of Life measured by Generic Quality of Life at 24 months.
Health-Related Quality of Life at 6 months. | 6 months
  Health-Related Quality of Life measured by Administration of QOL Measures at 6 months.
Health-Related Quality of Life at 12 months. | 12 months
  Health-Related Quality of Life measured by Administration of QOL Measures at 12 months.
Health-Related Quality of Life at 18 months. | 18 months
  Health-Related Quality of Life measured by Administration of QOL Measures at 18 months.
Health-Related Quality of Life at 24 months. | 24 months
  Health-Related Quality of Life measured by Administration of QOL Measures at 24 months.
Treatment Failures that are Not PTS. | 6-24 months
  Treatment Failures that are Not PTS (defined as one or more of the following during the 24 months post randomization: 1) the patient underwent an unplanned endovascular or surgical intervention for the treatment of severe symptomatic venous disease in the index leg within the first 24 months after randomization (2) the subject underwent an amputation in the index leg anytime within 24 months after randomization; or (3) the subject developed venous gangrene in the index leg within the first 24 months after randomization.
Severity of presenting DVT Symptoms at 6 months | 6 months
  Severity of presenting DVT Symptoms (Leg pain severity measured by pain scale) at 6 months
Severity of presenting DVT Symptoms at 12 months | 12 months
  Severity of presenting DVT Symptoms (Leg pain severity measured by pain scale) at 12 months
Severity of presenting DVT Symptoms at 18 months | 18 months
  Severity of presenting DVT Symptoms (Leg pain severity measured by pain scale) at 18 months
Severity of presenting DVT Symptoms at 24 months | 24 months
  Severity of presenting DVT Symptoms (Leg pain severity measured by pain scale) at 24 months
Severity of presenting DVT Symptoms at 6 months | 6 months
  Severity of presenting DVT Symptoms (Leg swelling measured by measuring calf swelling) at 6 months
Severity of presenting DVT Symptoms at 12 months | 12 months
  Severity of presenting DVT Symptoms (Leg swelling measured by measuring calf swelling) at 12 months
Severity of presenting DVT Symptoms at 18 months | 18 months
  Severity of presenting DVT Symptoms (Leg swelling measured by measuring calf swelling) at 18 months
Severity of presenting DVT Symptoms at 24 months | 24 months
  Severity of presenting DVT Symptoms (Leg swelling measured by measuring calf swelling) at 24 months
Degree of Resolution of Thrombus with PCDT at 6 months. | 6 months
  Degree of Resolution of Thrombus with PCDT (Assessed by two sets of venograms in PCDT arm, one baseline venogram of the proximal veins (popliteal vein through infrarenal IVC) obtained after initial catheter insertion into the venous system before PCDT; and one the final venogram of the proximal veins obtained after PCDT and any adjunctive procedures, before sheath removal. Marder score will be used to quantify clot burden. Marder score range 0-24, with 0 representing no thrombus and 24 representing complete thrombosis). The degree of thrombus elimination (% change in pre-PCDT and post-PCDT Marder score) will be calculated.
Degree of Resolution of Thrombus with PCDT at 12 months. | 12 months
  Degree of Resolution of Thrombus with PCDT (Assessed by two sets of venograms in PCDT arm, one baseline venogram of the proximal veins (popliteal vein through infrarenal IVC) obtained after initial catheter insertion into the venous system before PCDT; and one the final venogram of the proximal veins obtained after PCDT and any adjunctive procedures, before sheath removal. Marder score will be used to quantify clot burden. Marder score range 0-24, with 0 representing no thrombus and 24 representing complete thrombosis). The degree of thrombus elimination (% change in pre-PCDT and post-PCDT Marder score) will be calculated.
Degree of Resolution of Thrombus with PCDT at 18 months. | 18 months
  Degree of Resolution of Thrombus with PCDT (Assessed by two sets of venograms in PCDT arm, one baseline venogram of the proximal veins (popliteal vein through infrarenal IVC) obtained after initial catheter insertion into the venous system before PCDT; and one the final venogram of the proximal veins obtained after PCDT and any adjunctive procedures, before sheath removal. Marder score will be used to quantify clot burden. Marder score range 0-24, with 0 representing no thrombus and 24 representing complete thrombosis). The degree of thrombus elimination (% change in pre-PCDT and post-PCDT Marder score) will be calculated.
Degree of Resolution of Thrombus with PCDT at 24 months. | 24 months
  Degree of Resolution of Thrombus with PCDT (Assessed by two sets of venograms in PCDT arm, one baseline venogram of the proximal veins (popliteal vein through infrarenal IVC) obtained after initial catheter insertion into the venous system before PCDT; and one the final venogram of the proximal veins obtained after PCDT and any adjunctive procedures, before sheath removal. Marder score will be used to quantify clot burden. Marder score range 0-24, with 0 representing no thrombus and 24 representing complete thrombosis). The degree of thrombus elimination (% change in pre-PCDT and post-PCDT Marder score) will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Ehab A Eltahawy, MD, Principal Investigator — University of Toledo Health Science Campus
Locations (1):
- University of Toledo Medical Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vedantham S. Valvular dysfunction and venous obstruction in the post-thrombotic syndrome. Thromb Res. 2009;123 Suppl 4:S62-5. doi: 10.1016/S0049-3848(09)70146-X. PMID 19303507
- [Background] DUTCH CAVA-trial: CAtheter Versus Anticoagulation Alone for Acute Primary (Ilio)Femoral DVT. Clinicaltrial.gov
- [Result] Ashrani AA, Heit JA. Incidence and cost burden of post-thrombotic syndrome. J Thromb Thrombolysis. 2009 Nov;28(4):465-76. doi: 10.1007/s11239-009-0309-3. Epub 2009 Feb 18. PMID 19224134
- [Result] Kahn SR, Shrier I, Julian JA, Ducruet T, Arsenault L, Miron MJ, Roussin A, Desmarais S, Joyal F, Kassis J, Solymoss S, Desjardins L, Lamping DL, Johri M, Ginsberg JS. Determinants and time course of the postthrombotic syndrome after acute deep venous thrombosis. Ann Intern Med. 2008 Nov 18;149(10):698-707. doi: 10.7326/0003-4819-149-10-200811180-00004. PMID 19017588
- [Result] Kahn SR, Comerota AJ, Cushman M, Evans NS, Ginsberg JS, Goldenberg NA, Gupta DK, Prandoni P, Vedantham S, Walsh ME, Weitz JI; American Heart Association Council on Peripheral Vascular Disease, Council on Clinical Cardiology, and Council on Cardiovascular and Stroke Nursing. The postthrombotic syndrome: evidence-based prevention, diagnosis, and treatment strategies: a scientific statement from the American Heart Association. Circulation. 2014 Oct 28;130(18):1636-61. doi: 10.1161/CIR.0000000000000130. Epub 2014 Sep 22. No abstract available. PMID 25246013
- [Result] Comerota AJ, Grewal N, Martinez JT, Chen JT, Disalle R, Andrews L, Sepanski D, Assi Z. Postthrombotic morbidity correlates with residual thrombus following catheter-directed thrombolysis for iliofemoral deep vein thrombosis. J Vasc Surg. 2012 Mar;55(3):768-73. doi: 10.1016/j.jvs.2011.10.032. Epub 2012 Jan 24. PMID 22277690
- [Result] Schweizer J, Kirch W, Koch R, Elix H, Hellner G, Forkmann L, Graf A. Short- and long-term results after thrombolytic treatment of deep venous thrombosis. J Am Coll Cardiol. 2000 Oct;36(4):1336-43. doi: 10.1016/s0735-1097(00)00863-9. PMID 11028492
- [Result] Goldhaber SZ, Buring JE, Lipnick RJ, Hennekens CH. Pooled analyses of randomized trials of streptokinase and heparin in phlebographically documented acute deep venous thrombosis. Am J Med. 1984 Mar;76(3):393-7. doi: 10.1016/0002-9343(84)90656-9. PMID 6367454
- [Result] Elsharawy M, Elzayat E. Early results of thrombolysis vs anticoagulation in iliofemoral venous thrombosis. A randomised clinical trial. Eur J Vasc Endovasc Surg. 2002 Sep;24(3):209-14. doi: 10.1053/ejvs.2002.1665. PMID 12217281
- [Result] Bashir R, Zack CJ, Zhao H, Comerota AJ, Bove AA. Comparative outcomes of catheter-directed thrombolysis plus anticoagulation vs anticoagulation alone to treat lower-extremity proximal deep vein thrombosis. JAMA Intern Med. 2014 Sep;174(9):1494-501. doi: 10.1001/jamainternmed.2014.3415. PMID 25047081
- [Result] Enden T, Haig Y, Klow NE, Slagsvold CE, Sandvik L, Ghanima W, Hafsahl G, Holme PA, Holmen LO, Njaastad AM, Sandbaek G, Sandset PM; CaVenT Study Group. Long-term outcome after additional catheter-directed thrombolysis versus standard treatment for acute iliofemoral deep vein thrombosis (the CaVenT study): a randomised controlled trial. Lancet. 2012 Jan 7;379(9810):31-8. doi: 10.1016/S0140-6736(11)61753-4. Epub 2011 Dec 13. PMID 22172244
- [Result] Haig Y, Enden T, Grotta O, Klow NE, Slagsvold CE, Ghanima W, Sandvik L, Hafsahl G, Holme PA, Holmen LO, Njaaastad AM, Sandbaek G, Sandset PM; CaVenT Study Group. Post-thrombotic syndrome after catheter-directed thrombolysis for deep vein thrombosis (CaVenT): 5-year follow-up results of an open-label, randomised controlled trial. Lancet Haematol. 2016 Feb;3(2):e64-71. doi: 10.1016/S2352-3026(15)00248-3. Epub 2016 Jan 6. PMID 26853645
- [Result] Vedantham S, Goldhaber SZ, Julian JA, Kahn SR, Jaff MR, Cohen DJ, Magnuson E, Razavi MK, Comerota AJ, Gornik HL, Murphy TP, Lewis L, Duncan JR, Nieters P, Derfler MC, Filion M, Gu CS, Kee S, Schneider J, Saad N, Blinder M, Moll S, Sacks D, Lin J, Rundback J, Garcia M, Razdan R, VanderWoude E, Marques V, Kearon C; ATTRACT Trial Investigators. Pharmacomechanical Catheter-Directed Thrombolysis for Deep-Vein Thrombosis. N Engl J Med. 2017 Dec 7;377(23):2240-2252. doi: 10.1056/NEJMoa1615066. PMID 29211671
- See also: DUTCH CAVA-trial: CAtheter Versus Anticoagulation Alone for Acute Primary (Ilio)Femoral DVT. (NL28394) — https://clinicaltrials.gov/ct2/show/NCT00970619